CLINICAL TRIAL: NCT01613417
Title: Phase IV, Double-blind, Multi-center, Randomized, Crossover Study to Compare 0.1 mmol/kg of Prohance® With 0.1 mmol/kg of Gadovist®/Gadavist™ in Magnetic Resonance Imaging (MRI) of the Brain (TRUTH)
Brief Title: Comparison of Prohance® With Gadovist®/Gadavist™ in Magnetic Resonance Imaging (MRI) of the Brain
Acronym: TRUTH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: PH-107
Record Dates: First submitted 2012-06-04; First posted 2012-06-07 (Estimated); Results first posted 2015-06-03 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Brain Disease
Keywords: Have confirmed or are highly suspected of brain disease
MeSH Terms: conditions — Brain Diseases | interventions — gadoteridol; gadobutrol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MRI with Gadoteridol (Active Comparator): MRI after 0.1 mmol/kg IV ProHance, then with 0.1 mmol/kg Gadovist/Gadavist. MRI performed after both agents with identical sequences.
  Interventions: Drug: gadoteridol; Drug: gadobutrol
- MRI with Gadobutrol (Active Comparator): MRI after 0.1 mmol/kg IV Gadovist/Gadavist, then with 0.1 mmol/kg ProHance. MRI performed after both agents with identical sequences.
  Interventions: Drug: gadoteridol; Drug: gadobutrol

INTERVENTIONS:
Drug: gadoteridol — ProHance 0.1 mmol/kg
  Other Names: ProHance
Drug: gadobutrol — Gadovist/Gadavist 0.1 mmol/kg
  Other Names: Gadovist, Gadavist

SUMMARY:
This study aims at a direct comparison between ProHance (0.1 mmol/kg) and a validated comparator Gadovist/Gadavist (0.1 mmol/kg) in a crossover intra-individual design in subjects with brain tumors to confirm the identical overall technical and diagnostic performance of the two MR contrast agents.

DETAILED DESCRIPTION:
Adult patients were given two MRI exams, one after injection of ProHance (0.1 mmol/kg) and one after injection of Gadovist/Gadavist (0.1 mmol/kg). The exams were performed with identical equipment and imaging parameters with the order of the two exams randomized and 2-14 days between the first and the second MRI exam. Image data was evaluated by 3 expert neuroradiologist blinded to the agent administered and patient clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Are scheduled to undergo MRI
* Are willing to undergo two MRI procedures within 14 days
* Have confirmed or are highly suspected of brain disease likely to enhance as determined by the following:
* Clinical/neurological symptomatology;
* Diagnostic testing, such as CT or previous MRI examinations; or
* Have had previous brain surgery and are to be evaluated for recurrence.

Exclusion Criteria:

* Are pregnant or lactating females. Exclude the possibility of pregnancy:
* by testing on site at the institution within 24 hours prior to the start of each investigational product administration; or
* by history (i.e., tubal ligation or hysterectomy); or
* post menopausal with a minimum of 1 year without menses
* Have any known allergy to one or more of the ingredients in the investigational products, or have a history of hypersensitivity to any metals
* Have congestive heart failure (class IV according to the classification of the New York Heart Association; see Appendix A)
* Have suffered a stroke within a year
* Have received or are scheduled to receive any other contrast medium in the 24 hours preceding through the 24 hours following Exam 1, and in the 24 hours preceding through the 24 hours following Exam 2
* Have received or are scheduled to receive an investigational compound and/or medical device within 30 days before admission into the present study, through the 24 hours post-administration of the second investigational product.
* Have moderate-to-severe renal impairment, defined as a GFR/eGFR < 45 mL/min.
* Have been previously entered into this study
* Have received or are scheduled for one of the following:
* Surgery within three weeks prior to the first examination or between the two examinations
* Initiation of steroid therapy between the two examinations
* Radiosurgery between the two examinations
* Have any contraindications to MRI such as a pace-maker, magnetic material (i.e., surgical clips) or any other conditions that would preclude proximity to a strong magnetic field.
* Are suffering from severe claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2012-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gianpaolo Pirovano, MD, Study Director — Bracco Diagnostics, Inc
Locations (1):
- Holy Name Medical Center, Teaneck, New Jersey, United States

REFERENCES:
- [Result] Maravilla KR, Smith MP, Vymazal J, Goyal M, Herman M, Baima JJ, Babbel R, Vaneckova M, Zizka J, Colosimo C, Urbanczyk-Zawadzka M, Mechl M, Bag AK, Bastianello S, Bueltmann E, Hirai T, Frattini T, Kirchin MA, Pirovano G. Are there differences between macrocyclic gadolinium contrast agents for brain tumor imaging? Results of a multicenter intraindividual crossover comparison of gadobutrol with gadoteridol (the TRUTH study). AJNR Am J Neuroradiol. 2015 Jan;36(1):14-23. doi: 10.3174/ajnr.A4154. Epub 2014 Oct 9. PMID 25300984

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 229 patients were recruited from September 2012 through November 2013 at 19 clinical trial sites. Off-site assessment of the images was performed between 21 January and 3 April 2014 by 3 board-certified neuroradiologists blinded as to which contrast agent was used, patient clinical information, and the results of other imaging studies.
Pre-assignment Details: 229 patients were enrolled and signed informed consent. Each enrolled patient was randomized and dosed with at least one contrast agent.
Groups:
- Sequence 1 (ProHance Then Gadovist/Gadavist): Patients randomized to receive ProHance first
- Sequence 2 (Gadovist/Gadavist Then ProHance): Patients randomized to receive Gadovist/Gadavist first
Period: First Injection
Arm/Group | Sequence 1 (ProHance Then Gadovist/Gadavist) | Sequence 2 (Gadovist/Gadavist Then ProHance)
Started | 113 | 116
Completed | 113 | 116
Not Completed | 0 | 0
Period: Washout (no Second Injection/MRI)
Arm/Group | Sequence 1 (ProHance Then Gadovist/Gadavist) | Sequence 2 (Gadovist/Gadavist Then ProHance)
Started | 113 | 116
Completed | 100 | 109
Not Completed | 13 | 7
Not completed — Withdrawal by Subject | 13 | 7
Period: Second Injection
Arm/Group | Sequence 1 (ProHance Then Gadovist/Gadavist) | Sequence 2 (Gadovist/Gadavist Then ProHance)
Started | 100 | 109
Completed | 100 | 109
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Per Protocol
Groups:
- ProHance Then Gadovist/Gadavist; Gadovist/Gadavist Then ProHance: Per Protocol=patients who completed both exams, had global paired image data available, and had no major protocol violations
- Total: Total of all reporting groups
Arm/Group | ProHance Then Gadovist/Gadavist | Gadovist/Gadavist Then ProHance | Total
Number analyzed (Participants) | 93 | 105 | 198
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 70 | 140
  >=65 years | 23 | 35 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (14.27) | 55.9 (14.29) | 55.2 (14.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 58 | 108
  Male | 43 | 47 | 90
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 88 | 102 | 190
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 46 | 46 | 92
  Europe | 39 | 51 | 90
  Canada | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Global Diagnostic Preference Between the Two Exams
Description: Assessed by 3 blinded readers for each of the 198 patients who had post-dose exams for both ProHance and Gadovist/Gadavist. Readers assessed whether images with ProHance were preferred or images with Gadovist/Gadavist were preferred, or whether images after both exams were considered equal.
Time Frame: Comparison of image sets obtained within 2 to 14 days
Population: Per Protocol=patients who completed both exams, had global paired image data available, and had no major protocol violations
Measure: Number; unit: participant exams
Units Other Than Participants: Patient Exams
Groups:
- Reader 1: Paired exams reviewed by Reader 1
- Reader 2: Paired exams reviewed by Reader 2
- Reader 3: Paired exams reviewed by Reader 3
Arm/Group | Reader 1 | Reader 2 | Reader 3
Number analyzed (Participants) | 198 | 194 | 196
Number analyzed (Patient Exams) | 198 | 194 | 196
participant exams
  ProHance Preferred | 14 | 7 | 1
  Contrast Agents Equal | 171 | 180 | 195
  Gadovist/Gadavist Preferred | 13 | 7 | 0
Statistical Analysis 1: Comparison: Reader 1; Test type: Non-Inferiority or Equivalence — Power calculation was based on primary endpoint. 185 patients were deemed necessary for the lower limit of the observed 2-sided 95% confidence interval for the difference to exceed -5% with 85% power; p = 0.8516, Wilcoxon (Mann-Whitney) — P-value from Wilcoxon signed-rank test; Percentage PH better minus GV better = 0.5, 95% CI 2-sided [-4.6 to 5.6] — Difference in percentage ProHance better minus percentage Gadovist/Gadavist better (%)
Statistical Analysis 2: Comparison: Reader 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 1.0, Wilcoxon (Mann-Whitney) — P-value from Wilcoxon signed-rank test; Percentage PH better minus GV better = 0, 95% CI 2-sided [-3.8 to 3.8] — Difference in percentage ProHance better minus percentage Gadovist/Gadavist better (%)
Statistical Analysis 3: Comparison: Reader 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 1.0, Wilcoxon (Mann-Whitney) — P-value from Wilcoxon signed-rank test; Percentage PH better minus GV better = 0.5, 95% CI 2-sided [-0.5 to 1.5] — Difference in percentage ProHance better minus percentage Gadovist/Gadavist better (%)

2. Secondary Outcome: Lesion Border Delineation
Description: as for outcome 1
Time Frame: Comparison of image sets obtained within 2 to 14 days
Measure: Number; unit: participant exams
Units Other Than Participants: Patient Exams
Arm/Group | Reader 1 | Reader 2 | Reader 3
Number analyzed (Participants) | 198 | 194 | 196
Number analyzed (Patient Exams) | 198 | 194 | 196
participant exams
  ProHance Better | 8 | 2 | 1
  No Difference between Prohance and Gadovist/Gadavi | 181 | 189 | 195
  Gadovist/Gadavist Better | 9 | 3 | 0
Statistical Analysis 1: Comparison: Reader 1; Test type: Superiority or Other; p = 1.0, Wilcoxon (Mann-Whitney) — P-value from Wilcoxon signed-rank test
Statistical Analysis 2: Comparison: Reader 2; Test type: Superiority or Other; p = 1.0, Wilcoxon (Mann-Whitney) — P-value from Wilcoxon signed-rank test
Statistical Analysis 3: Comparison: Reader 3; Test type: Superiority or Other; p = 1.0, Wilcoxon (Mann-Whitney) — P-value from Wilcoxon signed-rank test

3. Secondary Outcome: Lesion Internal Morphology
Description: as for outcome 1
Time Frame: Comparison of image sets obtained within 2 to 14 days
Measure: Number; unit: participant exams
Units Other Than Participants: Patient Exams
Arm/Group | Reader 1 | Reader 2 | Reader 3
Number analyzed (Participants) | 198 | 198 | 198
Number analyzed (Patient Exams) | 198 | 194 | 196
participant exams
  ProHance better | 2 | 2 | 1
  No Difference Between ProHance and Gadovist/Gadavi | 195 | 188 | 195
  Gadovist/Gadavist betterB | 1 | 4 | 0
Statistical Analysis 1: Comparison: Reader 1; Test type: Superiority or Other; p = 1.0, Wilcoxon (Mann-Whitney) — P-value from Wilcoxon signed-rank test
Statistical Analysis 2: Comparison: Reader 2; Test type: Superiority or Other; p = 0.6875, Wilcoxon (Mann-Whitney) — P-value from Wilcoxon signed-rank test
Statistical Analysis 3: Comparison: Reader 3; Test type: Superiority or Other; p = 1.0, Wilcoxon (Mann-Whitney) — P-value from Wilcoxon signed-rank test

4. Secondary Outcome: Extent of Disease
Description: as for outcome 1
Time Frame: Comparison of image sets obtained within 2 to 14 days
Measure: Number; unit: participant exams
Units Other Than Participants: Patient Exams
Arm/Group | Reader 1 | Reader 2 | Reader 3
Number analyzed (Participants) | 198 | 198 | 198
Number analyzed (Patient Exams) | 198 | 194 | 196
participant exams
  ProHance Better | 1 | 2 | 1
  No Difference between ProHance and Gadovist/Gadavi | 196 | 190 | 195
  Gadovist/Gadavist Better | 1 | 2 | 0
Statistical Analysis 1: Comparison: Reader 1; Test type: Superiority or Other; p = 1.0, Wilcoxon (Mann-Whitney) — P-value from Wilcoxon signed-rank test
Statistical Analysis 2: Comparison: Reader 2; Test type: Superiority or Other; p = 1.0, Wilcoxon (Mann-Whitney) — P-value from Wilcoxon signed-rank test
Statistical Analysis 3: Comparison: Reader 3; Test type: Superiority or Other; p = 1.0, Wilcoxon (Mann-Whitney) — P-value from Wilcoxon signed-rank test

5. Secondary Outcome: Lesion Contrast Enhancement
Description: as for outcome 1
Time Frame: Comparison of image sets obtained within 2 to 14 days
Measure: Number; unit: participant exams
Units Other Than Participants: Patient Exams
Arm/Group | Reader 1 | Reader 2 | Reader 3
Number analyzed (Participants) | 198 | 198 | 198
Number analyzed (Patient Exams) | 198 | 194 | 196
participant exams
  ProHance Better | 14 | 10 | 2
  No Difference between ProHance and Gadovist/Gadavi | 170 | 174 | 193
  Gadovist/Gadavist Better | 14 | 10 | 1
Statistical Analysis 1: Comparison: Reader 1; Test type: Superiority or Other; p = 1.0, Wilcoxon (Mann-Whitney) — P-value from Wilcoxon signed-rank test
Statistical Analysis 2: Comparison: Reader 2; Test type: Superiority or Other; p = 1.0, Wilcoxon (Mann-Whitney) — P-value from Wilcoxon signed-rank test
Statistical Analysis 3: Comparison: Reader 3; Test type: Superiority or Other; p = 1.0, Wilcoxon (Mann-Whitney) — P-value from Wilcoxon signed-rank test

6. Secondary Outcome: Lesion to Background Ratio on Post T1-weighed Spin Echo Images
Description: Mean of difference in signal intensity postdose (ProHance - Gadovist/Gadavist)
Time Frame: 5-10 minutes Postdose
Population: Per-protocol population
Measure: Mean (Standard Deviation); unit: signal intensity
Units Other Than Participants: Lesions
Groups:
- Reader 1: Lesions reviewed by Reader 1
- Reader 2: Lesions reviewed by Reader 2
- Reader 3: Lesions reviewed by Reader 3
Arm/Group | Reader 1 | Reader 2 | Reader 3
Number analyzed (Participants) | 198 | 194 | 196
Number analyzed (Lesions) | 194 | 137 | 162
signal intensity | -0.02 (0.17) | -0.16 (1.12) | -0.01 (0.18)
Statistical Analysis 1: Comparison: Reader 1; Test type: Superiority or Other; p = 0.2758, Mixed Models Analysis; Mixed effect model with period, sequence, and IP and fixed effect and subject nested within sequence as random effect
Statistical Analysis 2: Comparison: Reader 2; Test type: Superiority or Other; p = 0.0676, Mixed Models Analysis; Mixed effect model with period, sequence, and IP and fixed effect and subject nested within sequence as random effect
Statistical Analysis 3: Comparison: Reader 3; Test type: Superiority or Other; p = 0.5267, Mixed Models Analysis; Mixed effect model with period, sequence, and IP and fixed effect and subject nested within sequence as random effect

7. Secondary Outcome: Percentage Signal Intensity Enhancement on Postdose Images
Description: Mean difference in percentage signal intensity enhancement on postdose T1-weighted SE/FSE images (ProHance - Gadovist/Gadavist)
Time Frame: 5-10 minutes Postdose
Population: Per-protocol population
Measure: Mean (Standard Deviation); unit: percentage signal intensity enhancement
Units Other Than Participants: Lesions
Arm/Group | Reader 1 | Reader 2 | Reader 3
Number analyzed (Participants) | 198 | 194 | 196
Number analyzed (Lesions) | 191 | 133 | 159
percentage signal intensity enhancement | 1.06 (28.61) | -2.09 (29.06) | -1.59 (29.16)
Statistical Analysis 1: Comparison: Reader 1; Test type: Superiority or Other; p = 0.6201, Mixed Models Analysis; Investigation product (IP) effect from mixed model with period, sequence, and IP as fixed effects and subject nested within sequence as random effect
Statistical Analysis 2: Comparison: Reader 2; Test type: Superiority or Other; p = 0.4514, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: Reader 3; Test type: Superiority or Other; p = 0.7722, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]

8. Secondary Outcome: Lesion Detection
Description: Lesion detection rate by contrast agent and reader
Time Frame: 5-10 minutes Postdose
Population: Per protocol patients with histologically confirmed lesions
Measure: Number; unit: participant exams
Groups:
- Reader 1 - ProHance; Reader 2 - ProHance; Reader 3 - ProHance: MRI after ProHance 0.1 mmol/kg
- Reader 1 - Gadovist/Gadavist; Reader 2 - Gadovist/Gadavist; Reader 3 - Gadovist/Gadavist: MRI after Gadovist/Gadavist 0.1 mmol/kg
Arm/Group | Reader 1 - ProHance | Reader 1 - Gadovist/Gadavist | Reader 2 - ProHance | Reader 2 - Gadovist/Gadavist | Reader 3 - ProHance | Reader 3 - Gadovist/Gadavist
Number analyzed (Participants) | 139 | 139 | 139 | 139 | 139 | 139
participant exams
  True Positive (Patients) | 133 | 135 | 137 | 136 | 136 | 132
  False Negative (Pa | 6 | 4 | 2 | 3 | 3 | 7
Statistical Analysis 1: Comparison: Reader 1 - ProHance vs Reader 1 - Gadovist/Gadavist; Test type: Superiority or Other; p = 0.3173, McNemar
Statistical Analysis 2: Comparison: Reader 2 - ProHance vs Reader 2 - Gadovist/Gadavist; Test type: Superiority or Other; p = 0.5637, McNemar
Statistical Analysis 3: Comparison: Reader 3 - ProHance vs Reader 3 - Gadovist/Gadavist; Test type: Superiority or Other; p = 0.0455, McNemar

9. Secondary Outcome: Accuracy for Tumor Characterization
Description: Blinded reader assessment of accuracy of tumor characterization (benign/malignant) - patient level assessment
Time Frame: 5-10 minutes Postdose
Population: Subjects with histologically confirmed lesions
Measure: Number; unit: participants
Arm/Group | Reader 1 - ProHance | Reader 1 - Gadovist/Gadavist | Reader 2 - ProHance | Reader 2 - Gadovist/Gadavist | Reader 3 - ProHance | Reader 3 - Gadovist/Gadavist
Number analyzed (Participants) | 128 | 128 | 128 | 128 | 128 | 128
participants
  Patients with Tumors Correctly Categorized | 94 | 96 | 106 | 101 | 93 | 83
  Patients with Tumors Incorrectly Categorized | 34 | 32 | 22 | 27 | 35 | 45
Statistical Analysis 1: Comparison: Reader 1 - ProHance vs Reader 1 - Gadovist/Gadavist; McNemar test of difference (ProHance minus Gadovist/Gadavist) in accuracy for tumor characterization; Test type: Superiority or Other; p = 0.6949, McNemar
Statistical Analysis 2: Comparison: Reader 2 - ProHance vs Reader 2 - Gadovist/Gadavist; McNemar test of difference (ProHance minus Gadovist/Gadavist) in accuracy for tumor characterization; Test type: Superiority or Other; p = 0.1317, McNemar
Statistical Analysis 3: Comparison: Reader 3 - ProHance vs Reader 3 - Gadovist/Gadavist; McNemar test of difference (ProHance minus Gadovist/Gadavist) in accuracy for tumor characterization; Test type: Superiority or Other; p = 0.0124, McNemar

ADVERSE EVENTS:
Time Frame: Up to 24 hours after contrast media injection
Description: All adverse events collected were categorized using MedDRA 16.1 and tabulated
Groups:
- Safety Population (ProHance): All enrolled patients who received a randomized injection of ProHance
- Safety Population (Gadovist/Gadavist): All enrolled patients who received a randomized injection of Gadovist/Gadavist
Arm/Group | Safety Population (ProHance) | Safety Population (Gadovist/Gadavist)
Serious Adverse Events (participants affected / at risk) | 0/222 | 0/216
Other Adverse Events (participants affected / at risk) | 15/222 | 8/216
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population (ProHance) (N=222) | Safety Population (Gadovist/Gadavist) (N=216)
Diarrhea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Fatigue (Gastrointestinal disorders) | 0 | 1
Feeling hot (General disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 4 | 1
Headache (Nervous system disorders) | 2 | 1
Lethargy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Orophanyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Vascular rupture (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Histologic confirmation of disease available for only 139/198 patients in the PP analysis. Of these, 128 patients had confirmed brain tumors and were available for the analyses of diagnostic performance (tumor detection and tumor characterization).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study results may be presented at scientific symposia or published in a peer-review journal after review by sponsor in accordance with the guidelines set forth in the applicable publication or financial agreement